CLINICAL TRIAL: NCT03831451
Title: Stroke Ready: A Stroke Preparedness Brief Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Lesli E. Skolarus, MD, Associate Professor of Neurology, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: U01MD010579-substudy; U01MD010579 (NIH)
Record Dates: First submitted 2019-01-24; First posted 2019-02-05 (Actual); Results first posted 2019-11-20 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Stroke
Keywords: stroke preparedness; behavioral intervention
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to a brief face-to-face stroke preparedness intervention compared to a healthy lifestyle stroke risk reduction intervention. After completing the outcome assessment, subjects will have the opportunity to receive the intervention that they were not initially randomized too.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stroke Preparedness Intervention (Experimental): The stroke preparedness educational intervention was designed with input from the community where it is being tested. It will be delivered in-person by a research team member. The intervention focuses on recognizing stroke symptoms and the importance of calling 911.
  Interventions: Behavioral: Stroke preparedness intervention
- Healthy lifestyle intervention (Active Comparator): The Healthy lifestyle stroke risk reduction educational intervention is based on patient materials from the American Heart Association. It will be delivered in-person by a research team member. The intervention focuses on stroke risk reduction.
  Interventions: Behavioral: Healthy lifestyle stroke risk reduction intervention

INTERVENTIONS:
Behavioral: Stroke preparedness intervention — Face-to-face interaction with research staff lasting between 5-10 minutes
  Arms: Stroke Preparedness Intervention
Behavioral: Healthy lifestyle stroke risk reduction intervention — Face-to-face interaction with research staff lasting between 5-10 minutes
  Arms: Healthy lifestyle intervention

SUMMARY:
This is a randomized controlled behavioral intervention trial to assess the efficacy of a brief intervention to increase stroke preparedness.

DETAILED DESCRIPTION:
This is a randomized controlled behavioral intervention trial to assess the efficacy of a brief intervention to increase stroke preparedness. Subjects will be randomized to a brief face-to-face stroke preparedness intervention compared to a healthy lifestyle stroke risk reduction intervention. The primary outcome is behavioral intent to call 911 using a self-administered survey

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2019-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lesli Skolarus, MD, MS, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Hamilton Community Health Network, Flint, Michigan
  - Hasselbring Senior Center, Flint, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Robles MC, Springer MV, Corches CL, Burke JF, Lin CC, Oliver A, Skolarus LE. Stroke Ready Very Brief Intervention Improves Immediate Postintervention Stroke Preparedness. Circ Cardiovasc Qual Outcomes. 2020 Dec;13(12):e006643. doi: 10.1161/CIRCOUTCOMES.120.006643. Epub 2020 Nov 26. No abstract available. PMID 33238728

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stroke Preparedness Intervention | Healthy Lifestyle Intervention
Started | 74 | 55
Completed | 74 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stroke Preparedness Intervention | Healthy Lifestyle Intervention | Total
Number analyzed (Participants) | 74 | 55 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (13) | 61 (15) | 61 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 33 | 79
  Male | 28 | 22 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 65 | 50 | 115
  White | 5 | 2 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Behavioral Intent to Call 911
Description: Change in Behavioral intent to call 911 using a self-administered survey. The survey is the Stroke Action test which was modified based on community input. Scores range from 0-12 for stroke. A higher score means greater stroke behavioral intent to call 911 for a stroke while a low score means lower behavioral intent to call 911 for a stroke.
Time Frame: Immediately (up to 10 minutes) before the brief intervention and then immediately (up to 10 minutes) after completing the brief intervention
Population: Mean changes from pre-intervention to post-intervention
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Stroke Preparedness Intervention | Healthy Lifestyle Intervention
Number analyzed (Participants) | 74 | 55
units on a scale | 2.1 (2.7) | 0.4 (2.2)

ADVERSE EVENTS:
Description: Adverse Events were not monitored/assessed.
Arm/Group | Stroke Preparedness Intervention | Healthy Lifestyle Intervention
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT03831451/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT03831451/ICF_001.pdf